CLINICAL TRIAL: NCT02431325
Title: A Study to Investigate Gastrointestinal Epithelial Integrity and Arterial Inflammation in Individuals With and Without HIV
Brief Title: A Study of the Gut Barrier and Blood Vessel Inflammation in Individuals With and Without HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ragon Institute of MGH, MIT and Harvard (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Janet Lo, MD, Assistant Professor in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P002669; 1R01HL123351-01 (NIH)
Record Dates: First submitted 2015-02-23; First posted 2015-05-01 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: HIV
Keywords: HIV; Atherosclerosis; Microbial Translocation; Teduglutide; Gastrointestinal Permeability; Inflammation
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teduglutide (Experimental): Teduglutide, subcutaneous injection, 0.05 mg/kg/day, 6 months duration
  Interventions: Drug: Teduglutide
- Placebo (Placebo Comparator): Placebo, subcutaneous injection, 6 months duration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teduglutide
  Other Names: Gattex
  Arms: Teduglutide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine whether teduglutide can repair a "leaky" gut, decrease inflammation, and prevent or treat plaque, a build-up of fat and other materials in the blood vessels of the heart, in people with HIV. HIV disease is linked to inflammatory changes and leakiness of the gut. These changes or conditions may increase the risk of developing heart and blood vessel disease. The investigators believe teduglutide can help repair the gut barrier in people with HIV, leading to a decrease in inflammation and plaque in the blood vessels of the heart.

DETAILED DESCRIPTION:
As more people with HIV gain access to combination antiretroviral therapy (cART), cardiovascular disease has become increasingly prevalent and a significant cause of mortality. Activation of the innate immune system may stimulate inflammatory mechanisms of atherosclerosis development. Loss of gastrointestinal (GI) mucosal epithelial integrity and loss of CD4+ T-lymphocytes in the intestinal lamina propria occur in HIV-infected patients and are not fully restored by cART. Translocation of microbial products from the intestinal lumen into the systemic circulation has been demonstrated to be increased in HIV-infected patients and the investigators hypothesize that it is a key driver of monocyte and macrophage activation. In turn, these pro-inflammatory monocytes and macrophages can induce atherosclerotic disease development. The purpose of the research study is to determine the effects of a glucagon-like peptide-2 analog, teduglutide, on intestinal epithelial integrity, microbial translocation across the gut lumen, markers of innate immune system activation including the monocyte transcriptome, bone, arterial inflammation, and atherosclerosis in a 6-month randomized, double-blind placebo-controlled proof of concept trial in HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 21-65 with previously diagnosed HIV disease
2. Stable anti-retroviral therapy (ART) as defined by no changes in ART regimen for >6 months
3. HIV viral load < 200 copies/mL
4. To be eligible for colonoscopy procedure, laboratory values that meet the following criteria:

   1. Hemoglobin > 9.0 g/dL
   2. Absolute neutrophil count ≥ 1000/mm3
   3. Platelet count ≥ 100,000/mm3
   4. Prothrombin time (PT) < 1.2 x upper limit of normal (ULN)
   5. Partial thromboplastin time (PTT) < 1.5 x ULN

4. Ability and willingness to give written informed consent and to comply with study requirements

Exclusion Criteria:

1. History of clinically significant gastrointestinal disease including but not limited to: colon cancer, intestinal obstruction, ulcerative colitis, Crohn's disease, or history of C. difficile within the past 3 months
2. First-degree relative with history of colon cancer
3. Active gall bladder, biliary or pancreatic disease
4. Female subject who is pregnant, nursing or less than 8 weeks post partum.
5. Use of any immunomodulatory agents within 30 days prior to study enrollment
6. History of intolerance, sensitivity, allergy or anaphylaxis to benzodiazepines or other narcotics to be used during the colonoscopy or upper endoscopy procedure
7. Contraindication to beta-blocker (including moderate to severe asthma or heart block) or nitroglycerin use as these drugs are given as part of the standard cardiac CT protocol. Previous allergic reaction to beta blocker or nitroglycerin.
8. Patients with previous allergic reactions to iodine-containing contrast media
9. Renal disease or creatinine >1.5 mg/dL (contrast will be administered during CT angiography of the heart)
10. History of requiring antibiotic prophylaxis for invasive procedures
11. History of myocardial infarction, decompensated cirrhosis, or any other condition that in the opinion of the investigator will compromise ability to participate in the study
12. Currently taking anticoagulants including but not limited to: heparin, warfarin (Coumadin), tinzaparin (Innohep), enoxaparin (Lovenox), danaparoid (Orgaran), dalteparin (Fragmin), clopidogrel (Plavix), prophylactic aspirin, and regular NSAID use
13. Subject taking any of the following medications: statins, systemic steroids (inhaled or nasal steroid therapy is permitted), interleukins, systemic interferons (e.g. local injection of interferon alpha for treatment of human papilloma virus is permitted), systemic chemotherapy including oral chemotherapeutic agents, methotrexate, octreotide, growth hormone, antiarrhythmics including digoxin, antiepileptics, immunosuppressants, vancomycin, rifampin, aminoglycosides, clonidine, prazosin, lithium and ritonavir-boosted lopinavir (Kaletra).
14. Subject has had two or more endoscopy procedures (sigmoidoscopy, upper endoscopy or colonoscopy) within the past 12 months for clinical purposes or other research studies.
15. Body weight greater than 300 lbs due to CT scanner table limitations
16. Active illicit drug use
17. Patients who report any significant radiation exposure over the course of the year prior to randomization. Significant exposure is defined as:

    1. More than 2 percutaneous coronary interventions (PCI) within 12 months of randomization
    2. More than 2 myocardial perfusion studies within the past 12 months
    3. More than 2 CT angiograms within the past 12 months
    4. Any subjects with history of radiation therapy
18. Patients already scheduled or being considered for a procedure or treatment

    1. requiring significant radiation exposure (e.g., radiation therapy, PCI, or catheter
    2. ablation of arrhythmia) within 12 months of randomization
19. History of malignancy
20. Prior recipient of a HIV vaccine

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12; Primary Completion 2020-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Lo, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Teduglutide: Teduglutide, subcutaneous injection, 0.05 mg/kg/day, 6 months duration
  Teduglutide
- Placebo: Placebo, subcutaneous injection, 6 months duration
  Placebo
Period: Overall Study
Arm/Group | Teduglutide | Placebo
Started | 17 | 15
Completed | 9 | 12
Not Completed | 8 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Declined to take study medication | 1 | 0
Not completed — Withdrew before starting study medication | 1 | 0
Not completed — Placebo shortage | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teduglutide | Placebo | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.3 [50.1 to 59.8] | 54.6 [49.5 to 59.2] | 56.1 [49.6 to 59.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 11 | 6 | 17
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Active Smoker [Count of Participants; unit: Participants] | 5 | 6 | 11
Current antiretroviral therapy (ART) use [Count of Participants; unit: Participants] | 17 | 15 | 32
Current non-nucleoside reverse transcriptase inhibitors (NNRTIs) use [Count of Participants; unit: Participants] | 3 | 5 | 8
Current protease inhibitor (PI) use [Count of Participants; unit: Participants] | 4 | 4 | 8
Current integrase strand transfer inhibitor (INSTI) use [Count of Participants; unit: Participants] | 13 | 9 | 22
CD4+ T-cell count [Mean (Standard Deviation); unit: cells/mm^3] | 639 (165) | 685 (225) | 660 (193)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (5.0) | 28.6 (4.4) | 27.8 (4.7)
Current statin use [Count of Participants; unit: Participants] | 7 | 4 | 11
HbA1c [Mean (Standard Deviation); unit: HbA1c, %] | 5.5 (0.4) | 5.6 (0.3) | 5.6 (0.3)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 180.82 (32.78) | 186.33 (35.04) | 183.41 (33.42)
Low density lipoprotein (LDL) cholesterol [Mean (Standard Deviation); unit: mg/dL] | 102.53 (27.93) | 113.93 (33.28) | 107.88 (30.60)
High density lipoprotein (HDL) cholesterol [Mean (Standard Deviation); unit: mg/dL] | 50.94 (16.54) | 48.33 (17.54) | 49.72 (16.79)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 136.59 (55.28) | 120.47 (42.93) | 129.03 (49.76)

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Target to Background Ratio of 18-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Uptake
Description: Change in maximum target to background ratio (TBRmax) of the most diseased segment (MDS) of the carotid index vessel. A negative number for the change in TBR implies a reduction in activity over time, which is considered an improvement in carotid arterial inflammation. Arterial FDG Uptake provides a measure of inflammation in the artery wall. TBR is target-to-background ratio (a measure of the ratio of the activity in the vessel wall divided by the blood background). The most diseased segment is the approximately 1-cm section of the vessel with the highest activity at baseline. The results are expressed as the change in the mean value, of the TBR, from baseline to 6 months.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with interpretable FDG-PET scans at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 5 | 10
ratio | -0.28 (0.29) | 0.01 (0.35)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.01, ANCOVA

2. Primary Outcome: Change in Intestinal Epithelial Integrity
Description: Change in plasma citrulline is calculated as log2 of the ratio of plasma citrulline at study end to baseline. Citrulline is a measure of functional small bowel mass, so a positive number is considered an improvement in intestinal epithelial integrity.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with available metabolite assessments at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: log2 ratio
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 10
log2 ratio | 0.39 (0.67) | -0.10 (0.22)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.04, t-test, 2 sided

3. Primary Outcome: Change in Soluble CD14 Concentration
Description: Soluble CD14 is a marker of monocyte activation. An increase in soluble CD14 concentration indicates an increase in inflammation.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with soluble CD14 available at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 10
ng/mL | 117.70 (387.56) | 142.85 (242.01)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.87, t-test, 2 sided

4. Secondary Outcome: Change in Intestinal CD4+ T-cells
Description: Change in CD161+CCR6+ (Th17) cells as a percentage of CD4+ T-cells in the duodenum. An increase in Th17 cells indicates a beneficial restoration of this CD4+ T-cell population in the small intestine, which are pathologically depleted in people with HIV.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with available biopsy samples from endoscopies at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T-cells
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 7 | 10
percentage of CD4+ T-cells | 13.17 (18.15) | -4.81 (15.98)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.047, t-test, 2 sided

5. Secondary Outcome: Change in CD14+CD86+CD40+ Monocytes
Description: Change in pro-inflammatory monocytes. A positive change indicates increased inflammation.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with peripheral blood flow cytometry data available at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention. Two participants in the placebo group did not have interpretable data for this monocyte population.
Measure: Mean (Standard Deviation); unit: percentage of CD14+ monocytes
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 7 | 8
percentage of CD14+ monocytes | -19.24 (14.12) | -3.31 (13.97)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided

6. Secondary Outcome: Change in HLA-DR+CD38+ CD8+ T Cells
Description: Change in activated CD8+ T Cells. A positive change indicates increased inflammation.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with peripheral blood flow cytometry at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: percentage of T Cells
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 7 | 10
percentage of T Cells | -0.33 (0.68) | 0.67 (1.22)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.07, t-test, 2 sided

7. Secondary Outcome: Change in HLA-DR+CD38+ CD4+ T Cells
Description: Change in activated CD4+ T Cells. A positive change indicates increased inflammation.
Time Frame: Change from baseline at 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of T Cells
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 7 | 10
percentage of T Cells | 0.0013 (0.19) | 0.058 (0.31)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.68, t-test, 2 sided

8. Secondary Outcome: Change in Soluble CD163 Concentration
Description: An increase in soluble CD163 concentration indicates an increase in inflammation.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with soluble CD163 data available at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 9
ng/mL | -9.26 (102.74) | 22.77 (85.95)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.49, t-test, 2 sided

9. Secondary Outcome: Change in Intestinal Fatty Acid Binding Protein Concentration
Description: An increase in I-FABP indicates an increase in intestinal mucosal damage.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with I-FABP data available at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 9
pg/mL | -270.04 [-675.05 to 1858.38] | -215.27 [-458.12 to 213.77]
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Plasma Riboflavin Concentration
Description: Change in plasma riboflavin is calculated as log2 of the ratio of plasma riboflavin at study end to baseline. A positive number indicates an increase in riboflavin levels.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with metabolite assessments at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: log2 ratio
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 10
log2 ratio | 0.55 (0.77) | -0.36 (0.89)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.04, t-test, 2 sided

11. Secondary Outcome: Change in Bone Mineral Density
Description: Change in femoral neck bone mineral density. An increase in bone mineral density is beneficial for bone health.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with bone density scans at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 6 | 10
g/cm^2 | 0.015 (0.021) | -0.0078 (0.022)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.07, t-test, 2 sided

12. Secondary Outcome: Change in Plaque Volume on Cardiac Computed Tomography Angiography
Description: Noncalcified plaque volume. Increased noncalcified plaque volume may indicate increased atherosclerosis.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with available cardiac CT data at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 6 | 10
mm^3 | -0.74 [-9.86 to 0.81] | 0.00 [-13.08 to 0.14]
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change in Hemoglobin A1c Percentage
Description: A higher hemoglobin A1c percentage indicates a higher blood glucose level over a 3 month average.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with HbA1c assessed at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Median (Inter-Quartile Range); unit: HbA1c, %
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 8 | 10
HbA1c, % | -0.1 [-0.1 to 0.2] | -0.1 [-0.3 to 0.0]
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change in Homeostatic Model Assessment-Insulin Resistance (HOMA-IR)
Description: A higher HOMA-IR indicates greater insulin resistance. Values greater than 2 suggests insulin resistance. HOMA-IR was calculated using a formula based on Matthews et al. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985;28(7):412-419.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with fasting glucose and fasting insulin assessed at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention and one participant in the active group that was not fasting for the study end blood draw.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 7 | 10
index | -0.40 (2.86) | 1.13 (3.20)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.33, t-test, 2 sided

15. Secondary Outcome: Change in Visceral Adipose Tissue (VAT) Area
Description: Abdominal VAT area was measured using single-slice abdominal CT at the level of the fourth lumbar vertebra. VAT is considered metabolically unhealthy fat.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with single-slice abdominal CT scans performed at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 6 | 10
cm^2 | -12.09 (46.59) | -7.94 (32.72)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.84, t-test, 2 sided

16. Secondary Outcome: Change in Subcutaneous Adipose Tissue (SAT) Area
Description: Abdominal SAT area was measured using single-slice abdominal CT at the level of the fourth lumbar vertebra.
Time Frame: Change from baseline at 6 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 6 | 10
cm^2 | -9.71 (39.91) | -0.11 (17.60)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.51, t-test, 2 sided

17. Secondary Outcome: Change in Body Mass Index (BMI)
Description: BMI is a measure of adiposity.
Time Frame: Change from baseline at 6 months
Population: The subset of participants with heights and weights measured at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 6 | 10
kg/m^2 | -0.33 (0.94) | -0.27 (1.14)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.93, t-test, 2 sided

18. Secondary Outcome: Change in Depressive Symptoms
Description: Change in the Center for Epidemiological Studies-Depression (CES-D) score. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Time Frame: Change from baseline at week 12 and at week 24
Population: The subset of participants with complete depression scales obtained by self-administered survey at baseline, 12 weeks, and 24 weeks, excluding one participant in the placebo group that discontinued ART during the intervention. Some participants that had depression scales at 24 weeks did not have them available at 12 weeks.
Measure: Median (Inter-Quartile Range); unit: CES-D score
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 7 | 11
CES-D score
  Change from baseline at week 24 | 1 [-3 to 3] | -3 [-6 to 0]
  Change from baseline at week 12: number analyzed (Participants) | 7 | 6
  Change from baseline at week 12 | 0 [-3 to 4] | 3 [-1 to 13]
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Change from baseline at week 24; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Teduglutide vs Placebo; Change from baseline at week 12; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change in Cognitive Performance, Defined as a Global Neurocognitive Z-score
Description: The Global Neurocognitive Z-Score is calculated as an average of the z-scores from the following neurocognitive assessments: Hopkins Verbal Learning Test (HVLT) Total Recall, HVLT Delayed Recall, HVLT Retention, HVLT Recognition, Wechsler Adult Intelligence Scale (WAIS) Digit Span Forward, WAIS Digit Span Backward, WAIS Digit Span Sequence, Stroop Word, Stroop Color, Stroop Color Word, Stroop Interference, Grooved Pegboard Dominant, and Grooved Pegboard Nondominant. A z-score of 0 corresponds with the population mean, and a positive z-score indicates better neurocognitive function than the population mean. A positive change indicates an improvement in neurocognitive function, and a negative change indicates a detriment to performance over time.
Time Frame: Change from baseline at week 24
Population: The subset of participants with neurocognitive testing results at baseline and study end, excluding one participant in the placebo group that discontinued ART during the intervention.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 5 | 9
z-score | 0.23 (0.39) | -0.04 (0.85)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.51, t-test, 2 sided

20. Secondary Outcome: Change in Domain-specific Cognitive Performance, Defined as a Domain-specific Neurocognitive Z-score
Description: Change in motor-specific performance z-score. A z-score of 0 corresponds with the population mean, and a positive z-score indicates better motor-specific performance than the population mean. A positive change indicates an improvement in motor-specific performance, and a negative change indicates a detriment to performance over time.
Time Frame: Change from baseline at week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 5 | 9
z-score | 1.73 (2.48) | -0.52 (1.72)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority; p = 0.07, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline, 6 months
Arm/Group | Teduglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 10/17 | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teduglutide (N=17) | Placebo (N=15)
Abdominal or epigastric pain, discomfort, cramping (Gastrointestinal disorders) | 5 | 3
Burping, gas (Gastrointestinal disorders) | 3 | 1
Bloating (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 4 | 2
Loose stool, diarrhea (Gastrointestinal disorders) | 2 | 4
Nausea, emesis (Gastrointestinal disorders) | 2 | 0
Decreased appetite (Gastrointestinal disorders) | 1 | 0
Viral gastroenteritis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Colonoscopy procedure-related adverse event (Gastrointestinal disorders) | 2 | 2
Emesis following IV contrast (Gastrointestinal disorders) | 0 | 1
Tubular adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Hyperplastic polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Sessile serrated polyp and polypoid of colonic mucosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bruising at injection site (Injury, poisoning and procedural complications) | 2 | 3
Bleeding at injection site (Injury, poisoning and procedural complications) | 0 | 1
Numbness at injection site (Injury, poisoning and procedural complications) | 0 | 1
Itching, burning at injection site (Injury, poisoning and procedural complications) | 0 | 1
Self-reported weight loss (Metabolism and nutrition disorders) | 1 | 0
Self-reported weight gain (Metabolism and nutrition disorders) | 0 | 3
Lightheadedness when taking the study drug and antiretroviral therapy together (General disorders) | 0 | 1
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02431325/Prot_SAP_000.pdf